CLINICAL TRIAL: NCT04927767
Title: A Self-controlled Clinical Trial on Denture Adhesives Used for Elderly Removable Denture Wearers
Brief Title: Denture Adhesives for Elderly Denture Wearers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-768
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Problem With Dentures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Denture adhesives (Experimental): Participants will be shown to apply the adhesive following the manufacturer's instructions. The denture is pressed firmly into place, then held firmly as the participant bites down to secure it. Participants will be instructed to apply the adhesive twice daily with an 8-hour interval.
  Interventions: Device: denture adhesive

INTERVENTIONS:
Device: denture adhesive — Denture adhesive is a commercially available denture care product used to adhere a denture to the oral mucosa, in order to improve the retention and stability.

SUMMARY:
Because of continuous change of the supporting oral tissues, removable dentures can gradually lose retention and stability, resulting in reduced masticatory efficiency. Denture adhesive is a commercially available material used to adhere a denture to the oral mucosa. Our previous review indicated that denture adhesive can improve denture retention, bite force and masticatory performance of complete denture wearers. However, related studies in partial dentures are rare. Therefore, this study aims to investigate the effects of denture adhesives on the masticatory performance and oral health related quality of life of removable partial denture and complete denture wearers.

Participants will be identified and recruited from the patient pool of the Prince Philip Dental Hospital (PPDH). Target patients are those who have problems with their existing dentures (for example, dissatisfied denture retention and stability, or reduced chewing efficiency), but do not plan to have new dentures. After sample size calculation, 47 participants are expected to be recruited for this clinical trial.

In this study, each participant will be interviewed by a trained interviewer and undergo a clinical examination. Information about the oral condition, denture condition, masticatory performance, oral health related quality of life, socio-demographic and other data will be recorded. Saliva samples will be collected for analysis of oral microorganisms.

A commercial copolymer-based cream adhesive (Polident, GlaxoSmithKline, Sussex, UK) is selected as the denture adhesive. Participants will be shown to apply the adhesive following the manufacturer's instructions. The denture is pressed firmly into place, then held firmly as the participant bites down to secure it. Participants will be instructed to apply the adhesive twice daily with an 8-hour interval.

Outcome measurements will be taken before application of denture adhesives, 1 week, 4 weeks and 12 weeks after usage of denture adhesives.

DETAILED DESCRIPTION:
In this study, each participant will be interviewed by a trained interviewer and undergo a clinical examination. Information about the oral condition, denture condition, masticatory performance, oral health related quality of life, socio-demographic and other data will be recorded. Saliva samples will be collected for analysis of oral microorganisms.

Details of the data collection methods are described below:

A. Oral condition

1. Oral mucosa moisture:

   A non-invasive oral moisture checking device (Mucus III, Life Co. Saitama, Japan) will be placed on the tongue and bilateral buccal mucosa of the participants to measure their oral moisture level (Murakami et al., 2009).
2. Dentition

   * Number and distribution of the remaining teeth and abutment teeth will be recorded.
   * Tooth mobility will be measured according to Miller's classification (Miller, 1938), and graded as follows:

     1. No detectable movement or only slight movement of the crown in horizontal direction (≤ 1mm)
     2. Visually increased mobility of the crown > 1 mm in a horizontal direction
     3. Severe mobility of the crown in both horizontal and vertical directions impinging on the function of the tooth.
   * DMFT (decayed, missing, and filled teeth) score will be computed for every individual. The tooth is recorded as D when dentine caries or cavity with or without fillings are present. The tooth is recorded as M when it has been. When a permanent or temporary filling is present, or when a filling is defective but not decayed, the tooth is counted as F.
   * The number and type of occluding pairs between upper and lower natural teeth and artificial teeth will be recorded.
3. Denture-bearing tissue Denture-bearing tissue will be clinically assessed according to Kapur's method (Kapur, 1967) with minor modification, in which the tissue is scored based on the ridge shape, tissue resiliency and depth of sulcus (location of border tissue attachment).
4. Condition of denture-bearing mucosal tissue

Presence of denture-related stomatitis will be recorded, which is characterised as inflammation and redness of the oral mucosa underneath the denture base. The Newton classification will be applied to classify the denture-related stomatitis (Scully, et al. 2008), which is as follows:

Type 1 - localized inflammation or pinpoint hyperemia; Type 2 - more diffuse erythema involving part or all of the mucosa which is covered by the denture; Type 3 - inflammatory nodular/papillary hyperplasia on the central hard palate or the alveolar ridge.

The determination will be based on the most severe segment of the edentulous region.

B. Denture condition

1. Denture base material and integrity Denture base material (acrylic or metal) will be recorded. Denture integrity will be assessed, and any of the following problems will be recorded: fracture of denture base or flange, broken clasps or rests, loss of abutment teeth, loss of non-abutment natural teeth, severe wear of prosthetic teeth, and others.
2. Denture retention and stability Denture retention and stability will be evaluated according to Kapur's, Corrigan's and Limpuangthip's methods (Kapur, 1967; Corrigan et al., 2002; Limpuangthip et al., 2018), and a sum score will be given to each denture.
3. Denture hygiene Denture hygiene will be determined by the Denture Cleanliness Index (Mylonas et al., 2014), which is scored from 0 to 4 according to the condition of staining, plaque, debris and calculus on denture.

   0 - Clean denture. No plaque is visibly seen, no staining, no plaque detectable.
   1. - Denture is visibly clean. Little staining (< 25% of fitting surface stained)
   2. - Denture has visible plaque and/or debris. Moderate staining of fit surface (25 - 50% of fitting surface stained)
   3. - Denture has visible plaque and/or debris. Severe staining of fit surface (> 50% of fitting surface stained)
   4. - Denture has visible calculus deposition, on any surface.

C. Masticatory performance

1. Maximum bite force:

   Maximum bite force in the incisal (central incisor) and bilateral posterior (first molar) regions will be measured by an occlusal force measurement device (iBite, Loadstar Sensors, CA, USA) (Fan et al., 2020). Two measurements will be taken for each site and the higher value will be recorded.
2. Masticatory efficiency:

   A colour-changeable chewing gum (XYLITOL, Lotte Co., Ltd., Saitama, Japan) will be applied to evaluate the masticatory efficiency of the participants. After 90 seconds of chewing, the chewed gum will be collected and the level of color change will be measured by a colorimeter (Shenzhen Threenh Technology Co., Ltd., Shenzhen, China). Three readings will be taken: at the centre and approximately 4 mm to its right and left, to obtain a mean a* value (CIE-L* a* b* colour system) (Fan et al., 2020).
3. Perceived chewing ability:

The validated Chinese version of the chewing function questionnaire (CFQ) that contains 10 food items in five levels of chewing difficulties with two food items in each level will be used (Fan et al., 2020). "No response" is given to the food item not consumed. The score of each food item will be summed to give a total CFQ score.

D. Oral health related quality of life:

The validated Chinese version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT-C) will be applied for assessing the OHRQoL of the participants (He et al., 2015). It consists of 19 items grouped into seven domains to describe the functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap of the participants, with higher score indicating lower OHRQoL.

E. Background information of denture wearers:

Demographic data including age and gender of the participants will be collected. Background information regarding denture wearing experience and habits, general satisfaction about the current dentures, number of currently using drugs will be also recorded.

Study design

This is a self-controlled clinical trial to investigate the influence of denture adhesives on the denture retention & stability, denture hygiene, masticatory performance and OHRQoL of elderly RPD wearers. The primary outcome is the change in masticatory performance. Ethics approval by the Institutional Review Board of the University of Hong Kong and Hospital Authority Hong Kong West Cluster has been obtained before implementation of the trial.

A commercial copolymer-based cream adhesive (Polident, GlaxoSmithKline, Sussex, UK) is selected as the denture adhesive. For participants in "both dentures group", the DA will be used for both dentures, while for participants in "single denture group", the DA will be used for eligible RPD only. Participants will be shown to apply the adhesive following the manufacturer's instructions. The denture is pressed firmly into place, then held firmly as the participant bites down to secure it. Participants will be instructed to apply the adhesive twice daily with an 8-hour interval.

Outcome measurements will be taken before application of denture adhesives, 1 week and 12 weeks after usage of denture adhesives. Phone calls will be given to the participants at 2 weeks, 4 weeks and 8 weeks after baseline to check their adherence and amount of denture adhesive used.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can communicate in Cantonese, Mandarin or English;
2. Subjects who wear either or both removable partial dentures (RPDs);
3. Subjects meet either one of the following criteria for extensive RPD: a. the corresponding arch has no posterior teeth (residual root will not be counted in) on one side or both sides; b. the corresponding arch has over half of the natural teeth missing (remaining teeth ≤ 8);
4. Participants with both upper and lower dentures meeting the requirement of "extensive RPD" will be included in "both dentures group", and participants with either upper or lower denture eligible will be included in "single denture group".

Exclusion Criteria:

1. Individuals who are unable to communicate clearly or having dementia;
2. Patients who are mostly bed-ridden, or suffering from infectious or life-threatening disease;
3. Individuals who are currently using denture adhesive;
4. Individuals who are allergic to denture adhesive;
5. Individuals whose denture is implant-supported or contraindicated for application of denture adhesive.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
masticatory efficiency | from baseline to 12-week follow-up
  A colour-changeable chewing gum (XYLITOL, Lotte Co., Ltd., Saitama, Japan) will be applied to evaluate the masticatory efficiency of the participants. After 90 seconds of chewing, the chewed gum will be collected and the level of color change will be measured in a 5-level visual scale (higher scale indicates better masticatory efficiency) and by a colorimeter (Shenzhen Threenh Technology Co., Ltd., Shenzhen, China). Three readings will be taken: at the centre and approximately 4 mm to its right and left, to obtain a mean a* value (CIE-L* a* b* colour system) (Fan et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Chiu Man Leung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- the University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No